CLINICAL TRIAL: NCT04310579
Title: Clinical Study to Investigate the Effect of the Combination of Psychotropic Drugs and an Opioid on Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other); Leiden University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SCR-009
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-11

CONDITIONS: Hypercapnia; Ventilatory Depression
Keywords: Opioids; Sedative psychotropic drugs
MeSH Terms: conditions — Hypercapnia; Respiratory Insufficiency | interventions — Oxycodone; Midazolam; Paroxetine; Quetiapine Fumarate

STUDY DESIGN:
Intervention Model Description: This clinical study consists of 3 parts:
  1. Up to 10 subjects in the Lead-In reproducibility assessment will have no drug treatment, only Read Rebreathing assessments.
  2. Approximately 20 subjects in Part 1 will be randomized to complete four treatments over four 1-day periods. Each period will be followed by 2 days of washout. Thus, Part 1 will have a cross-over component.
  3. Approximately 20 subjects in Part 2 will be randomized to complete three treatments over three 5-day periods. Each period will be followed by 7 days of washout. Thus, Part 2 will have a cross-over component.
  A maximum of 10 additional replacement subjects may be enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing. Subjects and staff will be blinded to treatment assignment. The blind will be maintained through a randomization schedule held by the dispensing pharmacist. Drugs will be over-encapsulated to maintain blinding during oral study drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lead-In (No Intervention): Read Rebreathing Reproducibility Assessment
- Part 1 Oxycodone and Midazolam (Active Comparator): In one period subjects receive oxycodone 10-15 mg immediate release (IR) tablets and intravenous (IV) placebo 1x per day.
  In a second period (randomized cross-over), subjects receive midazolam 0.0375-0.075 mg/kg IV and oral placebo tablet 1x per day.
  In a third period (randomized cross-over), subjects receive oxycodone 10-15 mg IR tablet and 0.0375-0.075 mg/kg midazolam IV 1x per day.
  In a fourth period (randomized cross-over), subjects receive oral placebo tablet and placebo IV 1x per day.
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
  Interventions: Drug: Oxycodone and Midazolam
- Part 2 Oxycodone, Paroxetine, and Quetiapine (Active Comparator): In one period, subjects receive: oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  In a second period (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  In a third period (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Interventions: Drug: Oxycodone, Paroxetine, and Quetiapine

INTERVENTIONS:
Drug: Oxycodone and Midazolam — In one period subjects receive oxycodone 10-15 mg immediate release (IR) and placebo IV 1x per day.
  In a second period (randomized cross-over), subjects receive midazolam 0.0375-0.075 mg/kg IV and oral placebo tablet 1x per day.
  In a third period (randomized cross-over), subjects receive oxycodone 10-15 mg IR tablet and 0.0375-0.075 mg/kg midazolam IV 1x per day.
  In a fourth period (randomized cross-over), subjects receive oral placebo tablet and placebo IV 1x per day.
  Arms: Part 1 Oxycodone and Midazolam
Drug: Oxycodone, Paroxetine, and Quetiapine — In one period, subjects receive: oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  In a second period (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  In a third period (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Arms: Part 2 Oxycodone, Paroxetine, and Quetiapine

SUMMARY:
Opioids can decrease breathing and co-administration of benzodiazepines with opioids can further decrease breathing. It is unknown whether certain other drugs also decrease breathing when co-administered with opioids. The objective of this study is to determine whether certain drugs combined with an opioid decrease breathing compared to breathing with an opioid alone.

In order to assess this, this study will utilize the Read Rebreathing method, where study participants breathe increased levels of oxygen and carbon dioxide. The increased levels of carbon dioxide cause the study participants to increase breathing. This increased breathing response can be decreased by opioids and benzodiazepines, and potentially other drugs. Using this procedure, low doses of opioids or benzodiazepines can be administered that have minimal-to-no effects on breathing when study participants are going about normal activities breathing room air, however breathing increases less than expected as carbon dioxide levels are increased. This study will also obtain quantitative pupillometry measurements before and after each rebreathing assessment to allow for comparisons of pupillary changes to ventilatory changes when subjects receive different drugs and drug combinations.

This study includes three parts: A Lead-In Reproducibility Phase and two main parts (Part 1 and Part 2). The Lead-In Reproducibility Phase will measure the variability between study participants and between repeated uses of the method in the same study participant within a day and between days. Part 1 will study an opioid alone, benzodiazepine alone, and their combination to show the methodology will detect changes in breathing at low doses of the drugs that are known to affect breathing. Part 2 will assess whether two drugs, selected due to their effects on breathing in a nonclinical model, decrease the breathing response when combined with an opioid compared to when an opioid is administered alone.

DETAILED DESCRIPTION:
Opioids can cause respiratory/ventilatory depression, and this can be exacerbated when opioids are co-administered with benzodiazepines. Research suggests this is caused by a reduced respiratory/ventilatory response to counteract increasing levels of systemic carbon dioxide (CO2). It is unknown whether certain other sedative psychotropic drugs can exacerbate opioid-induced respiratory/ventilatory depression. Studies were conducted to evaluate the effects of selected drugs in a non-clinical model. This clinical study will evaluate two drugs (quetiapine and paroxetine) that caused an effect when combined with oxycodone in the non-clinical model.

Study designs were evaluated that would allow a safe and controlled assessment of the effects of drug combinations on respiratory/ventilatory depression and a methodology was selected called the Read breathing procedure which introduces increased levels of CO2 to cause study participants to increase ventilation by having study participants rebreathe through a circuit with 93% oxygen (O2) and 7% CO2. Previous studies have shown this "hypercapnic ventilatory response" can be decreased by opioids and benzodiazepines and potentially other drugs. Using this procedure, low doses of opioids or benzodiazepines can be administered that have minimal-to-no effects on respiration/ventilation when study participants are going about normal activities breathing room air, however ventilation is decreased relative to the expected increase in ventilation as CO2 levels are increased during rebreathing. Thus, there is minimal risk of true respiratory depression (i.e. inadequate gas exchange) and, if needed, the investigators can immediately halt the experiment and have the study participant breathe room air or 100% O2.

Using the Read rebreathing methodology, the current clinical study was designed to generate data characterizing changes in the ventilatory response to hypercapnia when administering quetiapine and paroxetine alone or in combination with oxycodone. Information obtained from this study will inform on the potential for the specific studied drugs to affect ventilation when combined with an opioid and may also demonstrate the utility of this study design and methodology as an approach for evaluating the effect of an investigational drug and drug combinations on ventilatory depression. Thus, this study includes a lead-in reproducibility phase to quantify the intra- and inter-subject variability within a day and between days. In addition, this study includes a positive control phase with relatively low doses of opioid (oxycodone) alone, benzodiazepine (midazolam) alone and their combination to help assess assay sensitivity. While opioids and benzodiazepines have been studied alone and in combination with the rebreathing method previously, many of these studies are older and it is important to define the reproducibility and effects of the drugs at relatively low doses. Together, these components of the study will further define the reproducibility and sensitivity of the methodology that could be applied to a broader range of investigational drugs in the future to assess their safety when combined with opioids.

In addition, pupillary measurements have been used to study the pharmacodynamic effects of opioids and opioid antagonists (Skulberg et al, 2018; Rollins et al, 2014) and there has been interest in expanding its use in clinical studies. However, there are limited data directly comparing pupillary changes to ventilatory changes and some drugs may influence the pupillary response to opioids (Kummer et al, 2011). As an exploratory endpoint, this study will obtain quantitative pupillometry measurements before and after each rebreathing assessment to allow for comparisons of pupillary changes to ventilatory changes when subjects receive different drugs and drug combinations.

This study includes three parts: A Lead-In Reproducibility Phase and two main parts (Part 1 and Part 2). The lead-in reproducibility phase will quantify the intra- and inter-subject variability of the Read Rebreathing methodology within a day and between days. Part 1 is a positive control phase with doses of an opioid (oxycodone) alone, benzodiazepine (midazolam) alone, their combination, and placebo to help assess ability of the procedure to detect changes in ventilation. Part 2 will assess whether two sedative psychotropic drugs (quetiapine and paroxetine), selected due to their effects in a nonclinical model, decrease the ventilatory response to hypercapnia compared to an opioid (oxycodone) alone. The doses of oxycodone and midazolam were selected to be less than those previously administered in healthy volunteers undergoing the Read Rebreathing or similar respiratory circuit procedures that increase the inspired level of CO2. The doses of quetiapine and paroxetine were selected to reach clinical steady-state levels.

The Lead-In Reproducibility Phase will have up to 10 healthy volunteer participants enrolled in two cohorts of approximately five. Participants will perform the Read Rebreathing procedure five times on day 1 and five times on day 2.

Part 1 will be a 4-period randomized crossover study with approximately 20 healthy volunteer participants. Participants will receive four different treatments (oxycodone, midazolam, oxycodone + midazolam, and placebo) in a random order across each of the 1-day study periods. There will be two days of washout between each period. During each period, participants will perform the Read Rebreathing procedure seven times, for a total of 28 rebreathing assessments in Part 1. For Part 1, blood samples will also be collected for determination of study drug concentration.

Part 2 will be a 3-period randomized crossover study with approximately 20 healthy volunteer participants. Participants will receive three different treatments (oxycodone, oxycodone + quetiapine, and oxycodone + paroxetine) in a random order across each of the 5-day periods. Oxycodone will only be administered on day 1 and day 5 of each treatment period. The other drugs will be administered every day of the treatment period such that there will be lower concentrations on day 1 and higher concentrations on day 5, which are the days when oxycodone is co-administered. Read Rebreathing assessments will be performed on day 1 and day 5 to investigate the effect of paroxetine and quetiapine when combined with oxycodone compared to oxycodone alone. In addition, Read Rebreathing assessments will be performed on day 4 to determine the effect of paroxetine alone and quetiapine alone compared to placebo. There will be seven days of washout between each period. During each period, participants will perform the Read Rebreathing procedure 17 times, for a total of 51 rebreathing assessments in Part 2. For Part 2, blood samples will also be collected for determination of study drug concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 50 years of age, inclusive, who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at Screening and Check-in (Day -1).
5. Subject has no known or suspected allergies or sensitivities to any of the study drugs.
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the last application of study drug.
7. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the last application of study drug.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study

Exclusion Criteria:

1. Subject has history of opioid or psychotropic drug use within 60 days of the start of the study.
2. Subject has non-reactive or misshapen pupil(s) or damaged orbit structure or surrounding soft tissue is edematous or has an open lesion.
3. Subject has a Mallampati intubation score of >2 (for Part 1 and 2 only).
4. Subject Read Rebreathing data is of poor quality or subject does not agree to remain clean-shaven for all days when the Read Rebreathing procedure is being performed.
5. Subject has used any prescription or nonprescription drugs (including aspirin or [non-steroidal anti-inflammatory drugs] NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug. This includes prescription or nonprescription ophthalmic drugs.
6. Subjects are currently participating in another clinical study of an investigational drug or are have been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
7. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
8. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 h of dosing. Subjects must refrain from ingesting these throughout the study.
9. Subject has a history of sleep disorders, Panic Disorder, Panic Attacks, Generalized Anxiety Disorder, or any associated Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnosis or condition.
10. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study. This includes subjects with any underlying medical conditions that the Investigator believes would put subjects at increased risk of severe illness from COVID-19 based on the Centers for Disease Control and Prevention (CDC) guidelines. The CDC lists cancer, chronic kidney disease, chronic obstructive pulmonary disease, immunocompromised state from solid organ transplant, severe obesity, serious heart conditions, sickle cell disease, pregnancy, smoking and type 2 diabetes mellitus as conditions that put subjects at increased risk. Additionally, the CDC lists asthma (moderate-to-severe), cerebrovascular disease, cystic fibrosis, hypertension, immunocompromised state or immune deficiencies, neurologic conditions such as dementia, liver disease, pulmonary fibrosis, thalassemia, overweight, type 1 diabetes mellitus as conditions that might put subjects at increased risk.
11. Subject has any signs or symptoms that are consistent with COVID-19 per CDC recommendations. These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea may have COVID-19. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
12. Subject tests positive for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) by a molecular diagnostic test performed prior to admission.
13. Female subject is pregnant or lactating before enrollment in the study.
14. Subject has known or suspected allergies or sensitivities to any study drug.
15. Subject has clinical laboratory test results (hematology, serum chemistry) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
16. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
17. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
18. Subject has a history of or currently has hypoventilation syndrome or sleep apnea and is on non-invasive ventilation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as part of a manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as any eventual publications.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bailey PL, Andriano KP, Goldman M, Stanley TH, Pace NL. Variability of the respiratory response to diazepam. Anesthesiology. 1986 Apr;64(4):460-5. doi: 10.1097/00000542-198604000-00008. PMID 3083722
- [Background] Bourke DL, Warley A. The steady-state and rebreathing methods compared during morphine administration in humans. J Physiol. 1989 Dec;419:509-17. doi: 10.1113/jphysiol.1989.sp017883. PMID 2516128
- [Background] Cohen R, Finn H, Steen SN. Effect of diazepam and meperidine, alone and in combination, on respiratory response to carbon dioxide. Anesth Analg. 1969 May-Jun;48(3):353-5. No abstract available. PMID 5815096
- [Background] Forster A, Gardaz JP, Suter PM, Gemperle M. Respiratory depression by midazolam and diazepam. Anesthesiology. 1980 Dec;53(6):494-7. doi: 10.1097/00000542-198012000-00010. PMID 7457966
- [Background] Geddes DM, Rudolf M, Saunders KB. Effect of nitrazepam and flurazepam on the ventilatory response to carbon dioxide. Thorax. 1976 Oct;31(5):548-51. doi: 10.1136/thx.31.5.548. PMID 11571
- [Background] Ladd LA, Kam PC, Williams DB, Wright AW, Smith MT, Mather LE. Ventilatory responses of healthy subjects to intravenous combinations of morphine and oxycodone under imposed hypercapnic and hypoxaemic conditions. Br J Clin Pharmacol. 2005 May;59(5):524-35. doi: 10.1111/j.1365-2125.2005.02368.x. PMID 15842550
- [Background] Power SJ, Morgan M, Chakrabarti MK. Carbon dioxide response curves following midazolam and diazepam. Br J Anaesth. 1983 Sep;55(9):837-41. doi: 10.1093/bja/55.9.837. PMID 6137227
- [Background] Read DJ. A clinical method for assessing the ventilatory response to carbon dioxide. Australas Ann Med. 1967 Feb;16(1):20-32. doi: 10.1111/imj.1967.16.1.20. No abstract available. PMID 6032026
- [Background] Rebuck AS. Measurement of ventilatory response to CO2 by rebreathing. Chest. 1976 Jul;70(1 Suppl):118-21. doi: 10.1378/chest.70.1_supplement.118. No abstract available. PMID 939123
- [Background] Rigg JR. Ventilatory effects and plasma concentration of morphine in man. Br J Anaesth. 1978 Aug;50(8):759-65. doi: 10.1093/bja/50.8.759. PMID 678362
- [Background] Sarton E, Teppema L, Dahan A. Sex differences in morphine-induced ventilatory depression reside within the peripheral chemoreflex loop. Anesthesiology. 1999 May;90(5):1329-38. doi: 10.1097/00000542-199905000-00017. PMID 10319781
- [Background] van der Schrier R, Jonkman K, van Velzen M, Olofsen E, Drewes AM, Dahan A, Niesters M. An experimental study comparing the respiratory effects of tapentadol and oxycodone in healthy volunteers. Br J Anaesth. 2017 Dec 1;119(6):1169-1177. doi: 10.1093/bja/aex295. PMID 29029015
- [Background] van der Schrier R, Roozekrans M, Olofsen E, Aarts L, van Velzen M, de Jong M, Dahan A, Niesters M. Influence of Ethanol on Oxycodone-induced Respiratory Depression: A Dose-escalating Study in Young and Elderly Individuals. Anesthesiology. 2017 Mar;126(3):534-542. doi: 10.1097/ALN.0000000000001505. PMID 28170358
- [Background] Xu L, Chockalingam A, Stewart S, Shea K, Matta MK, Narayanasamy S, Pilli NR, Volpe DA, Weaver J, Zhu H, Davis MC, Rouse R. Developing an animal model to detect drug-drug interactions impacting drug-induced respiratory depression. Toxicol Rep. 2020 Jan 25;7:188-197. doi: 10.1016/j.toxrep.2020.01.008. eCollection 2020. PMID 32021808
- [Background] Kummer O, Hammann F, Moser C, Schaller O, Drewe J, Krahenbuhl S. Effect of the inhibition of CYP3A4 or CYP2D6 on the pharmacokinetics and pharmacodynamics of oxycodone. Eur J Clin Pharmacol. 2011 Jan;67(1):63-71. doi: 10.1007/s00228-010-0893-3. Epub 2010 Sep 21. PMID 20857093
- [Background] Rollins MD, Feiner JR, Lee JM, Shah S, Larson M. Pupillary effects of high-dose opioid quantified with infrared pupillometry. Anesthesiology. 2014 Nov;121(5):1037-44. doi: 10.1097/ALN.0000000000000384. PMID 25068603
- [Background] Skulberg AK, Tylleskar I, Nilsen T, Skarra S, Salvesen O, Sand T, Loftsson T, Dale O. Pharmacokinetics and -dynamics of intramuscular and intranasal naloxone: an explorative study in healthy volunteers. Eur J Clin Pharmacol. 2018 Jul;74(7):873-883. doi: 10.1007/s00228-018-2443-3. Epub 2018 Mar 22. PMID 29568976
- [Derived] Gershuny V, Florian J, van der Schrier R, Davis MC, Salcedo P, Wang C, Burkhart K, Prentice K, Shah A, Racz R, Patel V, Matta M, Ismaiel O, Boughner R, Ford KA, Rouse R, Stone M, Sanabria C, Dahan A, Strauss DG. Effect of midazolam co-administered with oxycodone on ventilation: a randomised clinical trial in healthy volunteers. Br J Anaesth. 2025 Apr;134(4):1170-1180. doi: 10.1016/j.bja.2024.11.047. Epub 2025 Feb 21. PMID 39986981
- [Derived] Florian J, van der Schrier R, Gershuny V, Davis MC, Wang C, Han X, Burkhart K, Prentice K, Shah A, Racz R, Patel V, Matta M, Ismaiel OA, Weaver J, Boughner R, Ford K, Rouse R, Stone M, Sanabria C, Dahan A, Strauss DG. Effect of Paroxetine or Quetiapine Combined With Oxycodone vs Oxycodone Alone on Ventilation During Hypercapnia: A Randomized Clinical Trial. JAMA. 2022 Oct 11;328(14):1405-1414. doi: 10.1001/jama.2022.17735. PMID 36219407

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Treatment Sequence ABCD: Participants first received treatment A and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment A: 10-15mg Immediate Release (IR) Oxycodone tablet + placebo IV Treatment B: Oral placebo + 0.0375-0.075 mg/kg midazolam IV Treatment C: 10-15 mg IR Oxycodone tablet + 0.0375-0.075 mg/kg midazolam IV Treatment D: Oral placebo + placebo IV
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
- Part 1 Treatment Sequence BDAC: Participants first received treatment B and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment B: Oral placebo + 0.0375-0.075 mg/kg midazolam IV Treatment D: Oral placebo + placebo IV Treatment A: 10-15mg Immediate Release (IR) Oxycodone tablet + placebo IV Treatment C: 10-15 mg IR Oxycodone tablet + 0.0375-0.075 mg/kg midazolam IV
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
- Part 1 Treatment Sequence CADB: Participants first received treatment C and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment C: 10-15 mg IR Oxycodone tablet + 0.0375-0.075 mg/kg midazolam IV Treatment A: 10-15mg Immediate Release (IR) Oxycodone tablet + placebo IV Treatment D: Oral placebo + placebo IV Treatment B: Oral placebo + 0.0375-0.075 mg/kg midazolam IV
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
- Part 1 Treatment Sequence DCBA: Participants first received treatment D and then crossed over to the sequential treatments with two days of washout in between treatments. Treatments are as follows:
  Treatment D: Oral placebo + placebo IV Treatment C: 10-15 mg IR Oxycodone tablet + 0.0375-0.075 mg/kg midazolam IV Treatment B: Oral placebo + 0.0375-0.075 mg/kg midazolam IV Treatment A: 10-15mg Immediate Release (IR) Oxycodone tablet + placebo IV
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
- Part 2 Treatment Sequence ABC: Participants first received treatment A and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
- Part 2 Treatment Sequence ACB: Participants first received treatment A and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
- Part 2 Treatment Sequence BAC: Participants first received treatment B and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
- Part 2 Treatment Sequence BCA: Participants first received treatment B and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
- Part 2 Treatment Sequence CAB: Participants first received treatment C and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
- Part 2 Treatment Sequence CBA: Participants first received treatment C and then crossed over to the sequential treatments with seven days of washout in between treatments. Treatments are as follows:
  Treatment C: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
  Treatment B: Subjects receive oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  Treatment A: Subjects receive oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
Period: Overall Study
Arm/Group | Lead-In | Part 1 Treatment Sequence ABCD | Part 1 Treatment Sequence BDAC | Part 1 Treatment Sequence CADB | Part 1 Treatment Sequence DCBA | Part 2 Treatment Sequence ABC | Part 2 Treatment Sequence ACB | Part 2 Treatment Sequence BAC | Part 2 Treatment Sequence BCA | Part 2 Treatment Sequence CAB | Part 2 Treatment Sequence CBA
Started | 10 | 5 | 5 | 5 | 5 | 4 | 5 | 3 | 4 | 4 | 5
Completed | 10 | 5 | 5 | 5 | 5 | 3 | 3 | 3 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive COVID-19 test | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Oxycodone and Midazolam: In one arm subjects receive oxycodone 10-15 mg immediate release (IR) tablets and intravenous (IV) placebo 1x per day.
  In a second arm (randomized cross-over), subjects receive midazolam 0.0375-0.075 mg/kg IV and oral placebo tablet 1x per day.
  In a third arm (randomized cross-over), subjects receive oxycodone 10-15 mg IR tablet and 0.0375-0.075 mg/kg midazolam IV 1x per day.
  In a fourth arm (randomized cross-over), subjects receive oral placebo tablet and placebo IV 1x per day.
  Note: Initial doses of oxycodone will be 10 mg, but may be increased to 15 mg if necessary based on criteria specified in protocol. Initial doses of midazolam will be 0.0375 mg/kg but may be increased to 0.075 mg/kg based on criteria specified in protocol.
- Part 2 Oxycodone, Paroxetine, and Quetiapine: In one arm, subjects receive: oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4.
  In a second arm (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4.
  In a third arm (randomized cross-over), subjects receive: oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5.
- Total: Total of all reporting groups
Arm/Group | Lead-In | Part 1 Oxycodone and Midazolam | Part 2 Oxycodone, Paroxetine, and Quetiapine | Total
Number analyzed (Participants) | 10 | 20 | 25 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [24 to 39] | 36 [32 to 41] | 35 [30 to 40] | 35 [30 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 11 | 24
  Male | 4 | 13 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 5 | 8
  Not Hispanic or Latino | 9 | 18 | 20 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 14 | 12 | 28
  White | 8 | 6 | 11 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 25 | 55
Body weight [Median (Inter-Quartile Range); unit: kg] | 77 [69 to 81] | 80 [74 to 89] | 68 [61 to 81] | 75 [65 to 83]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 25.6 [24.6 to 27.2] | 27.4 [24.9 to 28.3] | 24.8 [22.0 to 26.1] | 25.3 [24.0 to 27.8]

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Minute Ventilation at the 55 mm Hg End Tidal Carbon Dioxide (CO2) Point (VE55) on Day 1 for Oxycodone Combined With Midazolam and Oxycodone Alone.
Description: VE55 was estimated by analyzing rebreathing data using linear regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2). Rebreathing data were reviewed by 2 independent assessors blinded to study treatment and time of assessments to evaluate completeness of data for study outcomes. Resulting VE55 data of midazolam combined with oxycodone vs. oxycodone alone was compared using a linear mixed effects model with baseline VE55 as a continuous variable; treatment, sequence, and period as categorical variables; and participant as a random effect. R software was used for all analyses.
Time Frame: Part 1: 2 hour timepoint on treatment period Day 1
Population: All participants who finished more than 1 study period and completed rebreathing assessments at the 2-hour time point on day 1 were included in the primary analysis without imputation of missing data. One participant completed the study but did not have any completed rebreathing assessments at the 2-hour time point. Midazolam dose was escalated after the first five subjects, so those subjects who received the lower dose are excluded from summaries and comparison as specified in the protocol
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- Part 1: Oxycodone and Midazolam: Oxycodone 10 mg IR tablet and 0.075 mg/kg midazolam IV
- Part 1: Oxycodone: Oxycodone 10-15 mg immediate release (IR) tablets and intravenous (IV) placebo
Arm/Group | Part 1: Oxycodone and Midazolam | Part 1: Oxycodone
Number analyzed (Participants) | 14 | 19
L/min | 21.9 [17.1 to 26.6] | 24.1 [20.1 to 28.1]
Statistical Analysis 1: Comparison: Part 1: Oxycodone and Midazolam vs Part 1: Oxycodone; Part 1 is powered with consideration to both the effect of oxycodone versus placebo and oxycodone plus midazolam versus oxycodone. Assuming a -4 L/min effect size on VE55 and standard deviation of 5 L/min, there is greater than 90% power at a one-sided 0.05 significance level for a sample size of 20 subjects; Test type: Superiority; p = 0.22, Mixed Models Analysis — To demonstrate an effect of oxycodone with midazolam compared to oxycodone alone, it is necessary that the upper bound of the one-sided 95% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -2.2, 95% CI 1-sided [upper limit 2.5] — Comparison was the effect of oxycodone with midazolam compared to oxycodone alone

2. Primary Outcome: Part 2 - Minute Ventilation at the 55 mm Hg End Tidal Carbon Dioxide (CO2) Point (VE55) on Day 1 for Paroxetine or Quetiapine Combined With Oxycodone and Oxycodone Alone.
Description: VE55 was estimated by analyzing rebreathing data using linear regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2). Rebreathing data were reviewed by 2 independent assessors blinded to study treatment and time of assessments to evaluate completeness of data for study outcomes. Resulting VE55 data of paroxetine or quetiapine combined with oxycodone vs. oxycodone alone on Day 1 was compared using a linear mixed effects model with baseline VE55 as a continuous variable; treatment, sequence, and period as categorical variables; and participant as a random effect. R software was used for all analyses.
Time Frame: Part 2: 5 hour timepoint on Day 1
Population: All participants that completed paired rebreathing assessments with placebo-oxycodone and at least one of the other two study treatments (paroxetine-oxycodone or quetiapine-oxycodone combinations) for day 1 were included in the primary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- Part 2: Oxycodone + Placebo: Oxycodone 10-15 mg IR tablet 1x per day and oral placebo 3x per day on Days 1 and 5; and oral placebo 3x per day on Days 2-4
- Part 2: Oxycodone + Paroxetine: Oxycodone 10-15 mg IR tablet 1x per day, paroxetine 40 mg tablet 1x per day, and oral placebo 1x per day on Days 1 and 5; and paroxetine 40 mg tablet 1x per day and oral placebo 2x per day on Days 2-4
- Part 2: Oxycodone + Quetiapine: Oxycodone 10-15 mg IR tablet 1x per day, quetiapine 50 mg tablet 2x per day, and oral placebo 1x per day on Day 1; quetiapine 100 mg (2x50 mg tablets) 2x per day and oral placebo 1x per day on Day 2; quetiapine 150 mg (3x50 mg tablets) 2x per day and oral placebo 1x per day on Day 3; quetiapine 200 mg (4x50 mg tablets) 2x per day and oral placebo 1x per day on Day 4; and quetiapine 200 mg (4x50 mg tablets) 1x per day and oral placebo 1x per day on Day 5
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 20 | 20 | 20
L/min | 34.1 [31.1 to 37.2] | 29.2 [25.7 to 32.7] | 33.0 [30.0 to 36.0]
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; Sample size and power were calculated based on 2 primary outcomes (day 1 and day 5) with adjustment for multiplicity (α=.025). The assessments with paroxetine or quetiapine were considered as separate experiments. A sample size of 20 participants was determined to have 90 percent power at a 1-sided significance level to detect a 4 L/min decrease in the primary end point (ventilation at 55 mmHg end-tidal carbon dioxide) assuming a standard deviation of 5 L/min; Test type: Superiority; p = 0.01, Mixed Models Analysis — To demonstrate an effect of oxycodone with paroxetine compared to oxycodone alone, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -4.9, 97.5% CI 1-sided [upper limit -0.6] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.28, Mixed Models Analysis — To demonstrate an effect of oxycodone with quetiapine compared to oxycodone alone, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -1.2, 97.5% CI 1-sided [upper limit 2.8] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

3. Primary Outcome: Part 2 - Minute Ventilation at the 55 mm Hg End Tidal Carbon Dioxide (CO2) Point (VE55) on Day 5 for Paroxetine or Quetiapine Combined With Oxycodone and Oxycodone Alone.
Description: VE55 was estimated by analyzing rebreathing data using linear regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2). Rebreathing data were reviewed by 2 independent assessors blinded to study treatment and time of assessments to evaluate completeness of data for study outcomes. Resulting VE55 data of paroxetine or quetiapine combined with oxycodone vs. oxycodone alone on Day 5 was compared using a linear mixed effects model with baseline VE55 as a continuous variable; treatment, sequence, and period as categorical variables; and participant as a random effect. R software was used for all analyses.
Time Frame: Part 2: 5 hour timepoint on Day 5
Population: All participants that completed paired rebreathing assessments with placebo-oxycodone and at least one of the other two study treatments (paroxetine-oxycodone or quetiapine-oxycodone combinations) for day 5 were included in the primary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 19 | 19 | 19
L/min | 35.3 [31.4 to 39.2] | 25.1 [21.2 to 29.0] | 34.7 [30.9 to 38.5]
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -10.2, 97.5% CI 1-sided [upper limit -6.3] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -0.6, 97.5% CI 1-sided [upper limit 3.2] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

4. Secondary Outcome: Part 1 - Minute Ventilation at the 55 mm Hg End Tidal Carbon Dioxide (CO2) Point (VE55) for Oxycodone, Midazolam, and Placebo.
Description: VE55 was estimated by analyzing rebreathing data using linear regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2). Rebreathing data were reviewed by 2 independent assessors blinded to study treatment and time of assessments to evaluate completeness of data for study outcomes. Resulting VE55 data of oxycodone or midazolam alone compared to placebo was compared using a linear mixed effects model with baseline VE55 as a continuous variable; treatment, sequence, and period as categorical variables; and participant as a random effect. R software was used for all analyses.
Time Frame: Part 1: 2 hour timepoint on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- Part 1: Placebo: Oral placebo tablet and placebo IV
- Part 1: Midazolam: Midazolam 0.0375-0.075 mg/kg IV and oral placebo tablet
Arm/Group | Part 1: Placebo | Part 1: Midazolam | Part 1: Oxycodone
Number analyzed (Participants) | 19 | 14 | 19
L/min | 30.9 [26.9 to 34.8] | 30.0 [25.4 to 34.5] | 24.1 [20.1 to 28.1]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of oxycodone compared to placebo, it is necessary that the upper bound of the one-sided 95% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -6.8, 95% CI 1-sided [upper limit -2.5] — Comparison was the effect of oxycodone compared to placebo
Statistical Analysis 2: Comparison: Part 1: Midazolam vs Part 1: Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of midazolam compared to placebo, it is necessary that the upper bound of the one-sided 95% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -0.9, 95% CI 1-sided [upper limit 3.7] — Comparison was the effect of midazolam compared to placebo

5. Secondary Outcome: Part 2 - Minute Ventilation at the 55 mm Hg End Tidal Carbon Dioxide (CO2) Point (VE55) on Day 4 for Paroxetine, Quetiapine, and Placebo
Description: VE55 was estimated by analyzing rebreathing data using linear regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2). Rebreathing data were reviewed by 2 independent assessors blinded to study treatment and time of assessments to evaluate completeness of data for study outcomes. Resulting VE55 data of paroxetine, quetiapine, and placebo on Day 4 was compared using a linear mixed effects model with baseline VE55 as a continuous variable; treatment, sequence, and period as categorical variables; and participant as a random effect. R software was used for all analyses.
Time Frame: Part 2: 5 hour timepoint on Day 4
Population: All participants that completed paired rebreathing assessments with placebo-oxycodone and at least one of the other two study treatments (paroxetine-oxycodone or quetiapine-oxycodone combinations) for day 4 were included in the primary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 19 | 19 | 19
L/min | 41.7 [37.7 to 45.6] | 32.4 [28.2 to 36.5] | 42.8 [38.7 to 46.8]
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of paroxetine compared to placebo, it is necessary that the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -9.3, 97.5% CI 1-sided [upper limit -3.9] — Comparison was the effect of paroxetine compared to placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.67, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of quetiapine compared to placebo, it is necessary that the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = 1.1, 97.5% CI 1-sided [upper limit 6.4] — Comparison was the effect of quetiapine compared to placebo

6. Secondary Outcome: Part 1 - Maximum Observed Plasma Concentration (Cmax) of Oxycodone Alone vs. in Combination With Midazolam
Description: Cmax will be the maximum observed concentration for each treatment. Observations will be summarized using descriptive statistics.
Time Frame: Part 1: Day 1 at 0, 1, 2, 3, 4, 6, 8, 12, 24 hour
Population: The pharmacokinetic population will include all subjects who receive study drug and have at least 1 estimable PK parameter after dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Oxycodone and Midazolam | Part 1: Oxycodone
Number analyzed (Participants) | 20 | 20
ng/mL | 19.8 (27) | 21.8 (37)

7. Secondary Outcome: Part 2 - Cmax of Oxycodone Alone vs. in Combination With Paroxetine or Quetiapine on Day 1
Description: as for outcome 6
Time Frame: Part 2: Day 1 at 3, 4, 5, 6, 9, 12, 24 hour
Population: The pharmacokinetic population will include all subjects who receive study drug and have at least 1 estimable PK parameter on day 1 after dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 20 | 19 | 20
ng/mL | 18.3 (30) | 19.1 (25) | 22.9 (28)
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; Maximum oxycodone concentration was log-transformed and the values between study treatments were compared using a linear mixed effects model on day 1 with treatment as a categorical variable and participant as a random effect; Test type: Equivalence — A difference in exposure was concluded if the 2-sided 90% CI of the geometric mean ratio excluded 1, which is standard in pharmacokinetic studies; p = 0.33, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.06, 90% CI 2-sided [0.96 to 1.17] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.25, 90% CI 2-sided [1.14 to 1.37] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

8. Secondary Outcome: Part 2 - Cmax of Oxycodone Alone vs. in Combination With Paroxetine or Quetiapine on Day 5
Description: as for outcome 6
Time Frame: Part 2: Day 5 at 3, 4, 5, 6, 9, 12, 24 hour
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 19 | 19 | 19
ng/mL | 18.0 (26) | 23.4 (26) | 24.9 (26)
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; Maximum oxycodone concentration was log-transformed and the values between study treatments were compared using a linear mixed effects model on day 5 with treatment as a categorical variable and participant as a random effect; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.30, 90% CI 2-sided [1.19 to 1.43] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 8, analysis 1]; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.39, 90% CI 2-sided [1.22 to 1.57] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

9. Secondary Outcome: Part 1 - Area Under the Plasma Concentration-time Curve (AUC) of Oxycodone Alone vs. in Combination With Midazolam
Description: AUC will be calculated using noncompartmental methods for each treatment. Observations will be summarized using descriptive statistics.
Time Frame: Part 1: Day 1 at 0 (pre-dose), 1, 2, 3, 4, 6, 8, 12, 24 hour
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hour
Arm/Group | Part 1: Oxycodone and Midazolam | Part 1: Oxycodone
Number analyzed (Participants) | 20 | 20
ng/mL*hour | 129 (34) | 136 (38)

10. Secondary Outcome: Part 2 - AUC of Oxycodone Alone vs. in Combination With Paroxetine or Quetiapine on Day 1
Description: as for outcome 9
Time Frame: Part 2: Day 1 at 0 (pre-dose), 3, 4, 5, 6, 8, 9, 12, 24 hours
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 20 | 19 | 19
ng/mL*hr | 107 (25) | 107 (29) | 113 (25)
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; Area under the curve was log-transformed and the values between study treatments were compared using a linear mixed effects model on day 1 with treatment as a categorical variable and participant as a random effect; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.64, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.03, 90% CI 2-sided [0.91 to 1.17] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 10, analysis 1]; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.24, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.06, 90% CI 2-sided [0.98 to 1.15] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

11. Secondary Outcome: Part 2 - AUC of Oxycodone Alone vs. in Combination With Paroxetine or Quetiapine on Day 5
Description: as for outcome 9
Time Frame: Part 2: Day 5 on 0 (pre-dose), 3, 4, 5, 6, 8, 9, 12, 24 hours
Population: The pharmacokinetic population will include all subjects who receive study drug and have at least 1 estimable PK parameter on day 5 after dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
Number analyzed (Participants) | 19 | 19 | 19
ng/mL*hr | 102 (24) | 112 (30) | 129 (23)
Statistical Analysis 1: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Paroxetine; Area under the curve was log-transformed and the values between study treatments were compared using a linear mixed effects model on day 5 with treatment as a categorical variable and participant as a random effect; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.05, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.10, 90% CI 2-sided [1.02 to 1.19] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Part 2: Oxycodone + Placebo vs Part 2: Oxycodone + Quetiapine; [analysis description as in outcome 11, analysis 1]; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity; Geometric mean ratio = 1.27, 90% CI 2-sided [1.19 to 1.36] — Comparison was the effect of oxycodone and quetiapine compared to oxycodone and placebo

ADVERSE EVENTS:
Time Frame: Lead-in: 4 Days, Part 1: 11 Days, Part 2: 30 Days
Groups:
- Lead-In: Read Rebreathing Reproducibility Assessment (No intervention)
- Part 1: Placebo: Oral placebo + placebo IV (Part 1)
- Part 1: Midazolam: Oral placebo + midazolam IV (Part 1)
- Part 1: Oxycodone: Oxycodone + placebo IV (Part 1)
- Part 1: Oxycodone + Midazolam: Oxycodone + midazolam IV (Part 1)
- Part 2: Oxycodone + Placebo: Oxycodone + Placebo (Part 2)
- Part 2: Oxycodone + Paroxetine: Oxycodone + Paroxetine (Part 2)
- Part 2: Oxycodone + Quetiapine: Oxycodone + Quetiapine (Part 2)
Arm/Group | Lead-In | Part 1: Placebo | Part 1: Midazolam | Part 1: Oxycodone | Part 1: Oxycodone + Midazolam | Part 2: Oxycodone + Placebo | Part 2: Oxycodone + Paroxetine | Part 2: Oxycodone + Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20 | 0/20 | 0/20 | 0/20 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20 | 0/20 | 0/20 | 0/20 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/10 | 6/20 | 5/20 | 8/20 | 5/20 | 16/25 | 17/25 | 20/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (N=10) | Part 1: Placebo (N=20) | Part 1: Midazolam (N=20) | Part 1: Oxycodone (N=20) | Part 1: Oxycodone + Midazolam (N=20) | Part 2: Oxycodone + Placebo (N=25) | Part 2: Oxycodone + Paroxetine (N=25) | Part 2: Oxycodone + Quetiapine (N=25)
Pallor (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyparaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 8 (13) | 12 (16) | 3 (6)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 3 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 6 (7)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Medical device site irritation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 6 (7) | 7 (8)
Headache (Nervous system disorders) | 4 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 7 (9) | 7 (7) | 5 (5)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (6) | 7 (11)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04310579/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04310579/SAP_002.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04310579/ICF_000.pdf